CLINICAL TRIAL: NCT07082101
Title: Evaluating Biomarkers of Temporal Interference for Temporal Lobe Epilepsy Under SEEG
Brief Title: Temporal Interference for Temporal Lobe Epilepsy Under SEEG
Acronym: TITE-SEEG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252287
Record Dates: First submitted 2025-06-29; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporal interference (Experimental)
  Interventions: Other: temporal interference

INTERVENTIONS:
Other: temporal interference — In this intervertion, patients with SEEG operation will take temporal interference (TI) stimulation and the deep brain EEG will be monitorated through the entire experiment.

SUMMARY:
This study evaluates the effect of temporal interference (TI) stimulation on biomarkers in patients with temporal lobe epilepsy (TLE) under stereo-electroencephalography (SEEG), and provides theoretical basis for non-invasive TI treatment of temporal lobe epilepsy.

DETAILED DESCRIPTION:
10 patients aged 18-65 years with TLE assessed by semiology, video electroencephalogram and imaging in Epilepsy Center of Xijing Hospital (Xi'an, China) will be recruited. Clinical baseline data such as general information and history of seizures will be collected. The SEEG electrodes were implanted in the Department of neurosurgery of Xijing Hospital and after 24 hours TI will be performed with continuous SEEG monitoring. Finally, the biomarker changes of EEG signals before and after TI treatment were statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of drug refractory epilepsy and temporal lobe epilepsy;
* Patients undergoing SEEG;
* Able to cooperate the treatment and related inspection;
* Fully understands and signs informed consent.

Exclusion Criteria:

* Patients with temporal plus epilepsy;
* In status epilepticus;
* With other severe disease;
* Pregnancy or lactation women;
* Unable to tolerate SEEG or TI;
* At the same time to participate in other clinical trials;
* Withdraw consent procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of interictal electrophysiological biomaker changes in epilepsy | 24 hours after TI stimulation
  Electrophysiological biomarkers changes recorded by SEEG through the experiment.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China